CLINICAL TRIAL: NCT03396822
Title: Meningeal Inflammation on 7T MRI as a Tool for Measuring and Predicting Ocrelizumab Response in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Daniel Harrison, Associate Professor, University of Maryland, Baltimore
Other Study IDs: HP-00074320
Record Dates: First submitted 2018-01-04; First posted 2018-01-11 (Actual); Results first posted 2024-02-05 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; 7T MRI; Meningeal inflammation
MeSH Terms: conditions — Multiple Sclerosis | interventions — gadoteridol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Gadoteridol — gadolinium MRI contrast

SUMMARY:
Multiple Sclerosis (MS) is an autoimmune disorder of the central nervous system. In MS, inflammation is known to attack areas of the brain, spinal cord, and optic nerves; resulting in disability. Current MRI technology provides an adequate view of the impact of MS on the "white matter" of the brain, which contains many of the connections between neurons. Quantification of lesions in the white matter due to MS are a standard part of clinical trials and clinical care in MS. However, it has long been known that MS not only can affect the white matter, but also the "gray matter," which contains the majority of the nerve cells in the brain and can cause inflammation in the meninges (the protective tissue that surrounds the brain and spinal cord). Autopsy studies have shown that the inflammation seen in the meninges is driven by a B-cells, a subset of white blood cells and that meningeal inflammation may be responsible for damage to the gray matter of the brain.

Ocrelizumab is a new treatment for multiple sclerosis. This medication works by targeting and destroying circulating B-cells. It is thought that this may reduce the level of meningeal inflammation in patients with multiple sclerosis. By reducing meningeal inflammation, this medication may result in less damage to the gray matter and subsequently less disability in MS patients.

In this study, the investigators will evaluate the use of a method on 7 tesla (7T) MRI to identify inflammation in the meninges as a potential predictor of response to ocrelizumab treatment for multiple sclerosis. Further, the investigators will evaluate if this MRI technique can be used to monitor the long-term effect of the medication on meningeal inflammation and the development of damage to the gray matter of the brain.

DETAILED DESCRIPTION:
Twenty-two (22) participants will be recruited from the University of Maryland Center for Multiple Sclerosis Treatment and Research. Participants will be included if they are aged 18-65, have a diagnosis of relapsing or progressive multiple sclerosis per revised 2010 McDonald Criteria, and are planning to begin ocrelizumab therapy for multiple sclerosis, as prescribed by their treating physician. Participants will be excluded if they are unable to undergo an MRI due to metallic implants/devices or claustrophobia, have a history of allergy to gadolinium contrast, or are unable to provide informed consent.

All participants will undergo a baseline/screening study visit prior to initiation of ocrelizumab. This will include signing of informed consent, a clinical interview to collect demographic and clinical data, a physical examination to calculate the EDSS score, and implementation of the component tests of the Multiple Sclerosis Functional Composite (MSFC). All participants will then undergo an MRI on a 7T Philips Achieva scanner (housed at the Kennedy Krieger Institute, Baltimore, MD). This will be a whole brain MRI, including 0.7mm3 resolution magnetization prepared 2 rapid acquisition gradient echo (MP2RAGE) and MPFLAIR images acquired both pre- and post-intravenous infusion of gadolinium contrast.

MP2RAGE images will be processed to create T1 maps and T1-weighted images. All images (MPFLAIR included) will be co-registered to the pre-contrast MP2RAGE T1 map. Subtraction images will be created by subtracting the pre-contrast MPFLAIR scan from post-contrast images. Regions of hyperintensity on the subtraction image will be reviewed on anatomical images, and marked as regions of leptomeningeal enhancement if they have an amorphous appearance and are present in the leptomeningeal space.

Participants who are found to have leptomeningeal enhancement on their baseline scan will be considered as having passed screening and will proceed with further study procedures. Those that do not have meningeal enhancement on a baseline scan will not return for a follow up visit.

Participants who have passed screening (and thus have meningeal enhancement on their baseline scan) will then undergo initiation of ocrelizumab per clinical trial or commercial drug protocol as previously planned by their treating neurologists. Participants will then return for a follow up visit within 1 month after their 12 month ocrelizumab infusion. All of the above study procedures will be repeated on that date.

Follow up images for each subject will undergo co-registration to the pre-contrast MP2RAGE T1 map. This will allow co-registered review of baseline and 1 year follow up MPFLAIR images side-by-side for review of the presence or absence of enhancing foci noted at baseline on the 1 year follow up scan. Subtraction images will also be created utilizing the 1 year pre- and post-contrast MPFLAIR scan for quantification of the number of enhancing foci on the 1 year follow up scan by the same procedures as above. A semi-automated region growing painting tool will be used to create masks over areas of contrast enhancement, which will be used to quantify enhancing focus volume on the baseline and follow up scan. Further, subtraction mapping will be utilized to highlight regions of hypointensity present in the cortex on MP2RAGE T1 that were not present on baseline MP2RAGE T1, which would indicate a new cortical lesion at follow up.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of relapsing or primary progressive multiple sclerosis according to revised 2010 McDonald Criteria
* Ages 18 to 65, inclusive
* Have been prescribed ocrelizumab by their treating physician for treatment of multiple sclerosis, with the 1st infusion to occur within 30 days of enrollment

Exclusion Criteria:

* Inability to provide informed consent
* Inability to undergo MRI due to implantable devices or metallic foreign bodies considered unsafe in the MRI magnet
* Known severe allergic reaction (anaphylaxis) in the past to gadolinium contrast
* A current diagnosis of severe kidney failure and/or use of hemodialysis
* Currently pregnant or lactating
* History of a seizure disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with multiple sclerosis who have been prescribed ocrelizumab
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2023-05-25 (Actual); Study Completion 2023-05-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel M Harrison, M.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ocrelizumab Treated: Participants treated with ocrelizumab 600mg intravenous every 6 months
Period: Overall Study
Arm/Group | Ocrelizumab Treated
Started | 23
Completed | 14
Not Completed | 9
Not completed — No meningeal enhancement on baseline scan | 8
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- Participants With Baseline Meningeal Enhancement: Participants treated with ocrelizumab who had baseline meningeal enhancement
Arm/Group | Participants With Baseline Meningeal Enhancement
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.8 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 14
Meningeal enhancement on baseline scan [Count of Participants; unit: Participants] | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in the Number of Enhancing Leptomeningeal Foci on 1 Year Follow up Compared to Baseline in MS Patients Treated With Ocrelizumab.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: number of enhancing foci
Arm/Group | Participants With Baseline Meningeal Enhancement
Number analyzed (Participants) | 14
number of enhancing foci | 0.07 (2.9)

2. Secondary Outcome: Reduction in the Proportion of Participants With Meningeal Enhancement After Treatment With Ocrelizumab Compared to Pre-treatment Baseline.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With Baseline Meningeal Enhancement
Number analyzed (Participants) | 14
Participants | 8

3. Other Pre Specified Outcome: Change in the Volume of Contrast Enhancement on Follow up Compared to Baseline.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: mm3
Arm/Group | Participants With Baseline Meningeal Enhancement
Number analyzed (Participants) | 14
mm3 | -21.9 (77.6)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Participants With Baseline Meningeal Enhancement
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-12): https://cdn.clinicaltrials.gov/large-docs/22/NCT03396822/Prot_SAP_001.pdf